CLINICAL TRIAL: NCT04873856
Title: Multidimensional INDividualized NUTritional Therapy for Individuals with Severe Chronic Obstructive Pulmonary Disease
Brief Title: Multidimensional Individualized Nutritional Therapy for Individuals with Severe COPD
Acronym: MINDNUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Birgitte Lindegaard Madsen, Chief Physician, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MINDNUT NOH
Record Dates: First submitted 2021-04-23; First posted 2021-05-05 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Health-related quality of life; Nutrition; Mental health; Functional capacity; Anthropometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Psychological Well-Being | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intervention contains:
  1. individual nutritional plan
  2. regular contact
  3. friendly reminder/informal caregiver and
  4. weight dairy.
  Interventions: Dietary Supplement: Intervention
- Control Group (No Intervention): Standard of care

INTERVENTIONS:
Dietary Supplement: Intervention — The four dimensions of MINDNUT are described below:
  Nutritional plan: is conducted in collaboration with the participant based on nutritional registration and information about routines and habits to reach a daily protein target of 1.5 g/kg/day. The nutritional plan is adjusted at the regular contact, and nutritional supplementation will be handed out to the participant.
  Friendly reminder/informal caregiver: is a friendly reminder that encourage the participant to follow the nutritional plan and to ask for support (a note to hang on the refrigerator). The informal caregiver is a person with close contact to the participant.
  Regular contacts: The participant will be contacted on regular basis (with an interval of 7-14 days) via phone and besides nutritional plan, this conversation will be used to talk about well-being, compliance and potential side-effects.
  Weight diary: participants is instructed in keeping a weight diary which include registration of a daily weight.
  Arms: Intervention group

SUMMARY:
Individuals with severe chronic pulmonary disease often life isolated with a high burden of symptoms. Nutritional risk and low quality of life are common, and both associated with increased societal cost and poor prognosis. COPD is a complex and progressive disease with changing clinical states that influences nutritional status and quality of life in different ways. The primary aim is to improve quality of life for individuals with severe COPD.

120 individuals are recruited from the outpatient clinic at Nordsjællands Hospital in Denmark to a randomized controlled trial with two parallel groups (intervention and control). The intervention will last for 3 months comprising four elements including nutritional plan, regular contact, informal caregiver/friendly reminder and a weight dairy.

We expect that the intervention will improve quality of life, nutritional status and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 35 years
* Severe COPD defined as GOLD grade 2 group B or D OR GOLD grade 3 and 4 group ABCD
* Able to eat orally
* Live in own home
* Speak Danish or English
* Undernourished OR at risk of undernutrition defined as BMI ≤ 21 kg/m2 if < 70 years and BMI <22 kg/m2 if ≥70 years OR BMI 21-25 kg/m2 plus nutritional risk (nutritional risk screening score ≥3) if <70 years and BMI 22-25 kg/m2 plus nutritional risk if ≥70 years
* Stable phase

CHANGE: Undernourished OR at risk of undernutrition (a maximum BMI of 25 kg/m2) determined by Nutritional Risk Screening 2002 or Mini Nutritional Assessment Short Form according to the protocol published in Trials.

Exclusion Criteria:

* Active solid cancer" defined as cancer diagnosed within the previous six months, recurrent, regionally advanced, or metastatic cancer, cancer for which treatment had been administered within six months or hematological cancer that is not in complete remission
* Unable to sign informed consent e.g. due to severe dementia.
* Severe chronic renal failure defined as estimated glomerular filtration rate < 30 mL/min./1.73 m2 (ICD-10 codes N18.4 and N18.5
* Severe alcohol abuse (ICD-10 codes F10.2 and K70.x).

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 1 and 3 months after baseline
  Will be measured using the EQ-5D-5L

SECONDARY OUTCOMES:
Weight | 1 and 3 months after baseline
  Measured using an electronic scale (TANITA DC 430 SMA, TANITA, Denmark) to the nearest 0.1 kg
Body mass index | 1 and 3 months after baseline
  Calculated as weight (kg)/height (m2)
Hand grip strength | 1 and 3 months after baseline
  Measured using handdynanometer
Lower body strength | 1 and 3 months after baseline
  Measured using 30 second stand chair test
Number of unplanned acute hospitalizations | 1 and 3 months after baseline
  Obtained from patient files
Number of days in hospital | 1 and 3 months after baseline
  Obtained from patient files
Number of acute unplanned visits to emergency ward (<6 hours) | 1 and 3 months after baseline
  Obtained from patient files
Number of contacts to outpatient clinic (visits and phone calls) | up to 3 months after baseline
  Obtained from patient files
Disease specific quality of life | 1 and 3 months after baseline
  Obtained using COPD Assessment test (CAT). CAT contains 8 items with a scoring range of 0-40. The total score indicate the impact level COPD has on the everyday life ranging from low to very high. A total score of 5 is referred to the upper limit of normal in healthy non-smokers, a total score <10 indicate low impact, 10-20 indicate medium impact, whereas >20 and >30 indicate high and very high impact, respectively.
Mortality | up to 3 months after baseline
  will be obtained from patient files
Fat-free mass | 1 and 3 months after baseline
  Measured using bioelectrical impedance analysis
Fat mass | 1 and 3 months after baseline
  Measured using bioelectrical impedance analysis

OTHER OUTCOMES:
Total protein intake | 1 and 3 months after baseline
  Measured through 24-recall and calculated using MADlog (MADLOG, Denmark) in grams
Difference in protein requirement and protein intake | 1 and 3 months after baseline
  Intake measured through 24-recall and calculated using MADlog (MADLOG, Denmark) in grams adnd requirements is calculated as 1.5 g/kg/day.
Total energy intake | 1 and 3 months after baseline
  Measured through 24-recall and calculated using MADlog (MADLOG, Denmark) in kalories.
Difference in energy requirement and energy intake | 1 and 3 months after baseline
  Intake measured through 24-recall and calculated using MADlog (MADLOG, Denmark) in kalories. Requirements calculated as 30 kcal/kg/day if goal is weight maintenance and 45 kcal kg/day if goal is weight gain
Upper arm circumference | 1 and 3 months after baseline
  Measured using a measuring tape to the nearest 0.1 cm
Hip circumference | 1 and 3 months after baseline
  Measured using a measuring tape to the nearest 0.1 cm
Waist circumference | 1 and 3 months after baseline
  Measured using a measuring tape to the nearest 0.1 cm
Number of exacerbations | 1 and 3 months after baseline
  Obtained from patient files supplemented with self-reported information
Oxygen therapy | 1 and 3 months after baseline
  Self-reported. The participant is asked if he/she is currently using home oxygen.
Anxiety and depression | 1 and 3 months
  Measured using Hospital Anxiety and Depression Scale. The scale contains two subscales to evaluate risk of anxiety and depression. Each subscale contains 7 items with a total score from 0-21. Risk of anxiety and depression are based on a total score ≥8.
Physical activity (subjective) | 1 and 3 months after baseline
  Measured using the physical activity and vial signs questionnaire
Physical activity (objective) | 7 days from 1- months follow-up and 7 days from 3 months follow-up
  Measured using accelerometers (Activity AX3, Newcastle, United Kingdom)

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Lindegaard, MD, PhD, Principal Investigator — Department of Pulmonary and Infectious Diseases, Nordsjællands Hospital, 3400 Hillerød, Denmark
Locations (1):
- Nordsjællands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hegelund MH, Ritz C, Nielsen TL, Olsen MF, Soborg C, Braagaard L, Molgaard C, Krogh-Madsen R, Lindegaard B, Faurholt-Jepsen D. Multidimensional individualized nutritional therapy for individuals with severe chronic obstructive pulmonary disease: study protocol for a registry-based randomized controlled trial. Trials. 2023 Feb 6;24(1):86. doi: 10.1186/s13063-023-07099-1. PMID 36747276
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36747276/